CLINICAL TRIAL: NCT02226809
Title: Incidence of Residual Neuromuscular Block in Adult Patients in the Postanesthesia Care Unit. An Observational Cross-sectional Study of a Multicenter Cohort. The Residual Curarization in Spain Study (ReCuSS).
Brief Title: Multi-center Study of Residual Neuromuscular Block Incidence in the Post-anesthesia Care Unit
Acronym: ReCuSS
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Collaborators: General University Hospital of Valencia (Other); Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Carlos Luis Errando, MD, PhD, staff anesthesiologist, General University Hospital of Valencia
Other Study IDs: CEO-BNM-2014-01
Record Dates: First submitted 2014-08-20; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Incomplete Reversal of Neuromuscular Block; Postoperative Respiratory Complications
Keywords: Muscle relaxants; Postoperative complications, respiratory; General anesthesia; Postanesthesia care unit; Neuromuscular block reversal
MeSH Terms: conditions — Muscle Hypotonia; Postoperative Complications | interventions — Accelerometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General anesthesia: Evaluation of RNMB. Application of accelerometry to patients after general anesthesia receiving at least one intermediate action nondepolarizing neuromuscular blocking agent dose
  Interventions: Device: Accelerometry

INTERVENTIONS:
Device: Accelerometry — Application of TOF stimulus (40 mA, three to four times) and recording TOFr in the PACU
  Other Names: TOF-Watch

SUMMARY:
Residual neuromuscular block (RNMB) is frequent in the immediate postoperative period and is a source of complications, mainly respiratory. The incidence is variable due to multiple factors. In Spain the incidence is unknown.

The investigators hypothesize that a number of patients in the postanesthesia care unit (PACU) present with RNMB after general anesthesia using intermediate action neuromuscular block agents (NMBA).

The main objective is to know the incidence of RNMB in Spanish hospitals. Secondary objectives are to observe the possible relationship with other pre- and intraoperative factors.

DETAILED DESCRIPTION:
Residual neuromuscular block (RNMB) is frequent in the immediate postoperative period and is a source of complications, mainly respiratory. This includes recovery delay or hospital discharge delays, respiratory insufficiency or infections, unforeseen ICU admissions, and prolonged ICU stays.

The incidence is variable due to multiple factors. Age, gender, surgery, NMBA type and doses, temperature, medications, etc.

In several studies it has been found and incidence between 6-80%. Few studies have been focused in evaluating the incidence in the whole country, as representing a global anesthesia practice. In Spain the incidence is unknown.

The investigators hypothesize that a number of patients in the postanesthesia care unit (PACU) present with RNMB after general anesthesia using intermediate action NMBA.

The main objective is to know the incidence of RNMB in Spanish hospitals, by means of an observational cross-sectional multicenter study .

Secondary objectives are to observe the possible relationship with other pre- and intraoperative factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years-old
* General anesthesia with non-depolarizing NMBA
* Transferred extubated on spontaneous ventilation to the PACU

Exclusion Criteria:

* American Society of Anesthesiologists physical status IV-V
* emergency and cardiac surgery
* patients unable to respond adequately at the moment of pre- or postoperative evaluation (psychiatric diseases, excessive somnolence, agitation, etc.)
* noncompensated diabetes mellitus or diabetic neuropathy
* symptomatic severe hypothyroidism (or untreated), or scheduled for total thyroidectomy
* chronic or acute renal insufficiency
* severe hepatopathy (Child-Pugh B, C)
* intraoperative blood transfusion >3 blood units
* intraoperative maintained arterial hypotension
* arrival to the PACU intubated or with instrumented airway (including surgical)
* pre- or perioperative drugs intake affecting the neuromuscular transmission
* neuromuscular diseases affecting the physiology of the neuromuscular system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Residual neuromuscular block incidence (TOFr<0.9) measured by accelerometry in the PACU | Upon arrival to the PACU. Single evaluation.
  Patients operated on under general anesthesia including intermediate duration NMBA were evaluated by means of an accelerometer in the PACU immediately upon arrival. Train-of-four ratio (TOFr) is evaluated.
  The evaluator does'nt know the patient-related information, including intraoperative management.

SECONDARY OUTCOMES:
Respiratory or airway postoperative complications in the PACU | During PACU stay, an expected average of 4 hours
  Evaluation of respiratory complications or events in the PACU (asking the anesthesiologist in charge or PACU medical record) to discharge to the ward.

OTHER OUTCOMES:
Relationship of RNMB with preoperative patient related factors | Upon patients arrival to the PACU
  Analysis of the preoperative visit record and anesthesia record: ASA class, and patient's demographics and characteristics
Relationship of RNMB with intraoperative anesthesia-related factors | Upon PACU arrival
  anesthesiologist-in-charge experience, type of anesthesia, intraoperative drugs administered and doses, reversal drugs and doses.
Relationship of RNMB with surgery-related factors | Upon PACU arrival
  Relationship of RNMB with surgery related factors (surgical speciality, type of surgery -high risk vs low to intermedium risk, laparoscopic vs no laparoscopic-, duration), blood losses.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos L Errando, MD, PhD, Principal Investigator — Servicio de Anestesiologia. Consorcio Hospital General Universitario de Valencia; Ignacio Garutti, MD, PhD, Principal Investigator — Servicio de Anestesiologia. Hospital Universitario Gregorio Marañon
Locations (25):
- Spain (25):
  - Hospital General de Elda, Elda, Alicante
  - Hospital de Bellvitge, Badalona, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic Universitari, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General de Castellón, Castellon, Castellón
  - Complejo Hospitalario Universitario, A Coruña, Coruña
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital de Manacor, Manacor, Palma de Mallorca
  - Hospital Universitario Son Espases, Palma de Mallorca, Palma de Mallorca
  - Hospital Xeral de Vigo, Vigo, Pontevedra
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Universitario Dr Peset, Valencia, Valencia
  - Hospital Universitario Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Basurto, Basurto, Vizcaya
  - Hospital Miguel Servet, Zaragoza, Zaragoza